CLINICAL TRIAL: NCT04096339
Title: RECoVER: Reduction in Sedation: Colonoscopy vs Esophagoduodenoscopy First
Brief Title: Reduction in Sedation: Colonoscopy vs Esophagoduodenoscopy First
Acronym: RECoVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ala'a Sharara, MD, Professor of Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BIO-2018-0629
Record Dates: First submitted 2019-07-11; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia, Recovery
Keywords: Colonoscopy; EGD; Sedation; procedural sequence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGD followed by Colonoscopy (Active Comparator): Randomized to group Esophagogastroduodenoscopy followed by Colonoscopy
  Interventions: Other: EGD followed by Colonoscopy
- Colonoscopy followed by EGD (Active Comparator): Randomized to group Colonoscopy followed by Esophagogastroduodenoscopy
  Interventions: Other: Colonoscopy followed by EGD

INTERVENTIONS:
Other: Colonoscopy followed by EGD — Colonoscopy is done first followed by EGD
  Arms: Colonoscopy followed by EGD
Other: EGD followed by Colonoscopy — Esophagoduodenoscopy (EGD) is done first followed by Colonoscopy
  Arms: EGD followed by Colonoscopy

SUMMARY:
The purpose of this research is to compare the effect of different procedural sequences on the time to recovery and the propofol sedation requirements in patients undergoing bidirectional endoscopy with sedation.

The two sequences are:

* Colonoscopy followed by Esophagogastroduodenoscopy (EGD)
* EGD followed by Colonoscopy

DETAILED DESCRIPTION:
120 patients will be asked to participate in the trial. The subject will undergo both procedures in the order assigned by the randomization sheet. During the procedure, the endoscopist and anesthesiologists will collect data including but not limited to vital signs (heart rate, blood oxygen level, blood pressure) and level of sedation through the Bispectral Index Monitor (BIS). After completing the procedures, the patient will be approached in the recovery room by the study coordinator who will administer the Modified Post Anesthesia Discharge Scoring System (M-PADSS) scale every 5 minutes until a score of 9 or higher is obtained on two consecutive attempts. 24 hours following the procedure, the study coordinator will call the patient in order to assess the patient's cognitive function and drowsiness after they were discharged from the endoscopy unit.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Scheduled EGD and colonoscopy on the same day
* Scheduled to Anaesthesiologist administered sedation during the procedure

Exclusion Criteria:

* Age below 18
* Known allergy or adverse reaction to Propofol, Midazolam or opioid medication (ex: fentanyl)
* Medical contraindication to Anaesthesia
* Sleep apnea
* American Society of Anesthesiologists classification (ASA) >3
* Inpatient status
* Pregnant or lactating women
* Known cirrhosis
* Chronic Kidney Disease (stage 4 or 5)
* Known psychological disorder
* Known cognitive dysfunction
* Significant gastroparesis
* Gastric outlet obstruction
* Ileus
* Known or suspected bowel obstruction or perforation
* Having a stoma
* Compromised swallowing reflex or mental status
* Prior colon resection or gastric surgery
* Age above 75 years
* Chronic use of more than 1 psychoactive drug (Benzodiazepines, Tricyclic antidepressants, antipsychotics, selective serotonin receptor inhibitors, serotonin norepinephrine receptor inhibitors, Monoamine oxidase inhibitor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Time to discharge | 1 hour
  Time from end of procedures to patient discharge

SECONDARY OUTCOMES:
Propofol dose | 1 hour
  Propofol sedation requirements
Depth of anesthesia | 1 hour
  Bispectral Index (BIS) tracking of depth of anesthesia throughout the two procedures. BIS is a single dimensionless number generated by EEG analysis.
Cognitive impairment | 24 hours
  An assessment of cognitive impairment after the subject emerges from sedation, using the Modified Post Anesthesia Discharge System (M-PADS)
Adverse events during sedation | 1 hour
  apnea, desaturations, hypotension, bradycardia and other hemodynamical disturbances during sedation

CONTACTS AND LOCATIONS:
Overall Officials: Ala I Sharara, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut - Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Mokahal A, Daher HB, Yamout R, Hoshaimi N, Ayoub C, Shaib Y, Sharara AI. Randomized controlled trial of procedural sequence for same-day bidirectional endoscopy under monitored anesthesia care (RECoVER Trial). IGIE. 2023 Jul 25;2(3):282-291. doi: 10.1016/j.igie.2023.07.014. eCollection 2023 Sep. PMID 41646987